CLINICAL TRIAL: NCT05460468
Title: Adaptive Neuromodulation of Working Memory Networks in Aging and Dementia
Brief Title: Neuromodulation of Memory in Aging
Acronym: TMS-AD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: Pro00110872
Record Dates: First submitted 2022-06-06; First posted 2022-07-15 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Mild Cognitive Impairment; MCI
Keywords: TMS; Transcranial Magnetic Stimulation; Memory
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: The study has three Aims and thus three models.
  For Aim 1, the primary outcome measure is fMRI BOLD. Researchers will estimate the dose-response relationship between TMS intensity and BOLD response in two cortical sites for response to TMS.
  For Aim 2 the primary outcome measure is impact of closed-loop TMS treatment on working memory task performance.
  For Aim 3, the primary outcome measure is the strength of mediation of brain health (e.g., vascular density) predictors of cognition.
Who Masked: Participant
Masking Description: This is a within-subjects design, such that both active and sham stimulation (i.e., masking) trials will occur in all subjects.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- TMS-Randomized (Experimental): Three different closed-loop conditions will be tested, each triggered by the presence of a sustained period of alpha-band power. In the first condition, arrhythmic TMS trains with a stochastic (randomized) inter-pulse interval, will be used to disrupt cortical alpha oscillations and thus be expected to enhance memory performance.
  Interventions: Device: Transcranial Magnetic Stimulation
- TMS-Ordered (Experimental): Three different closed-loop conditions will be tested, each triggered by the presence of a sustained period of alpha-band power. In the second condition, rhythmic (ordered) alpha-frequency TMS trains, with the expectation that this alpha stimulation will further entrain a synchronization during the task and thereby worsen memory performance.
  Interventions: Device: Transcranial Magnetic Stimulation
- TMS-Sham (Sham Comparator): Three different closed-loop conditions will be tested, each triggered by the presence of a sustained period of alpha-band power. In a third condition, sham stimulation will be delivered at the same randomized inter-pulse interval, but with no TMS delivered to the brain.
  Interventions: Device: Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Transcranial Magnetic Stimulation — Transcranial magnetic stimulation (TMS) is a noninvasive procedure that uses magnetic fields to stimulate nerve cells in the brain to improve a variety of cognitive conditions, and to probe the dynamics of normal brain function.
  Other Names: TMS rTMS

SUMMARY:
The proposed research will use closed-loop transcranial magnetic stimulation (TMS) based on individualized brain networks to establish parameters that can reliably control brain states. This will be tested in healthy aging and mild cognitive impairment (MCI) cohorts. The investigators will study network activation and neural oscillatory mechanisms underlying the network that regulates working memory and then target this network using closed-loop TMS to the Prefrontal Cortex. Investigators will measure the impact of TMS on working memory performance and task-based neural activity. The project will use brain stimulation and network modeling techniques to enhance working memory in healthy older adults and MCI and will demonstrate the value of closed-loop, network-guided TMS for future clinical applications.

DETAILED DESCRIPTION:
Dementia due to Alzheimer's disease (AD) is a leading public health concern in the US with enormous care costs and no effective pharmacotherapy despite multiple clinical trials. Multiple studies have shown mild cognitive impairment (MCI) to be a precursor risk for AD and to be more amenable to intervention. While preclinical studies have shown that directly modulating activity in the prefrontal cortex (PFC) using non-invasive brain stimulation techniques, such as transcranial magnetic stimulation (TMS), can modulate cognitive function in healthy older adults, there is little evidence of reliable efficacy in MCI.

The investigators posit three reasons for this lack of efficacy. First, there is no established means of estimating a reliable biomarker and unique dose-response relationship between TMS intensity and brain activity. Second, standard TMS protocols fail to capture the dynamic nature of cognitive states and the reaction of endogenous brain states to exogenous neuromodulation. Third, no studies using TMS in AD-related populations have accounted for the influence of cerebrovascular disease in the response to TMS. The investigators propose to address these shortcomings by using closed-loop TMS, based on individualized brain networks to establish parameters that can reliably control brain states during normal memory functioning in healthy aging and MCI.

To achieve this goal, the investigators will study network activation and neural oscillatory mechanisms underlying the network that regulates working memory (WM), a cognition function with a reliable prefrontal cortex (PFC) network characterization. The investigators will then target this network using closed-loop TMS to the PFC and measure the impact on WM performance and task-based neural activity. This approach uses concurrent TMS-fMRI to identify dose-response relationships in the working memory network. Next, the investigators apply novel closed-loop TMS to perturb this network using temporally-precise TMS-EEG. Lastly, the investigators will integrate information collected via fMRI and EEG into a single computational framework to model spatiotemporal dynamics of the global brain network and predict the success of the TMS-related response in our MCI cohort. The project will use cutting-edge brain stimulation and network modeling techniques to enhance WM in healthy older adults and MCI and will provide a demonstration of the value of closed-loop, network-guided TMS for future clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Willing to provide consent

Exclusion Criteria:

* History of any Axis I DSM-V disorder, excluding major depressive disorder or generalized anxiety disorders
* Current history of substance abuse or dependence (excluding nicotine)
* Intracranial implants (e.g. aneurysms clips, shunts, stimulators, cochlear implants, or electrodes), cardiac pacemakers, or vagus Nerve stimulation device
* Increased risk of seizure for any reason, including prior diagnosis of epilepsy, seizure disorder, increased intracranial pressure, or history of significant head trauma with loss of consciousness for ≥ 5 minutes.
* Neurological disorder including, but not limited to: space occupying brain lesion; any history of seizures, history of cerebrovascular accident; fainting, cerebral aneurysm, Dementia, Hungtington chorea; Multiple Sclerosis.
* Current use of medications known to lower the seizure threshold and/or affect working memory

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-03-28 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Working Memory Task | Collected during TMS-EEG (Day 4)
  The difference in memory accuracy between TMS conditions (random vs. ordered vs. sham stimulation) on a working memory task. Each trial of the task consists of stimulus presentation of an array of letters, a delay period in which subjects alphabetize the letters, and probe period where subjects indicate whether the number corresponds to the alphabetized position of the letter probe presented. Memory is subsequently assessed as a function of TMS condition.
Functional network connectivity | Collected during the initial neuroimaging session (Day 2)
  Functional network connectivity/activity is estimated by comparing the hemodynamic time courses of two or more regions of the brain. The correlation between the time courses of each pair of regions is termed functional network connectivity. The Working Memory Network (WMN) is identified by comparing fMRI-based functional network connectivity for high vs low working memory load (e.g., remembering 4 versus 3 items).
Vascular density (VAD) | Collected during the second neuroimaging session (Day 3)
  This measure of neurovascular brain health, vascular density (VAD), as estimated by an automated method of segmenting veins with a magnetic resonance imaging (MRI) sequence known as susceptibility weighted imaging. This measure can be used to estimate the dilation of cerebral veins, and therefore VAD.
EEG-based connectivity | Collected during TMS-EEG (Day 4)
  EEG data will be source reconstructed to a fine-grained grid and timecourses of the solution points are averaged per region and per subject. The imaginary part of the coherence (iCoh) of averaged EEG source signals will be assessed within the alpha and theta frequency bands to build EEG-based connectivity matrices ("connectomes") for alpha- and theta-based connectivity, for each subject.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | Collected during the initial screening visit (Day 1)
  The MoCA was designed as a rapid screening instrument for mild cognitive dysfunction. This widespread tool is used to assesses different cognitive domains: attention and concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. The principle outcome measure is a summary score combining performance on each subtest. Scores range from 0 to 30. A higher score indicates intact cognitive functions.
National Institutes of Health (NIH) Toolbox Cognitive Battery | Collected during the initial screening visit (Day 1)
  The primary outcome measure of the NIH Toolbox is a Crystallized or Fluid Intelligence score. Fluid intelligence involves comprehension, reasoning and problem solving, while crystallized intelligence involves recalling stored knowledge and past experiences. These scores are normalized and scaled to reflect a 1-100 range. Higher scores indicate better performance.
Hopkins Verbal Learning Test (HVLT-2) | Collected during the initial screening visit (Day 1)
  The Hopkins Verbal Learning Test (HVLT-R) consists of memorization of a list of words to test the ability to recall immediately after memorization (immediate recall) and after a 20-minute delay (delayed recall). These scores are normalized to reflect a 1-100 percentile range. Higher scores indicate better performance.
Brief Visuospatial Memory Test (BVMT-R) | Collected during the initial screening visit (Day 1)
  The BVMT-R is a commonly used assessment tool to measure visuospatial learning and memory. A visual display of six simple figures arranged in a 2 × 3 matrix is shown to participants for three consecutive 10-second trials. Scoring of the immediate and delayed recall as well as copy trials are based on the accuracy of the drawings and the location of the figures. These scores are normalized to reflect a 1-100 percentile range. Higher scores indicate better performance.
Number Span Forwards/ Backwards | Collected during the initial screening visit (Day 1)
  Span tests measure the ability of a subject to remember a series of numbers in forward or reverse order. These scores are normalized to reflect a 1-100 percentile range. Higher scores indicate better performance.
Category & Phonemic Verbal Fluency | Collected during the initial screening visit (Day 1)
  Fluency tests measure the participant's ability to generate new exemplars for each categorical (e.g., farm animals) or phonemic (e.g., words starting with "b") prompts. The number of exemplars generated is recorded as the primary outcome for this test. These scores are normalized to reflect a 1-100 percentile range. Higher scores indicate better performance.
Trail Making Test | Collected during the initial screening visit (Day 1)
  The purpose of the "Trails" test is to gauge the ability of the participant to trace paths between a series of letters and numbers on a sheet of paper, and can provide insights into a person's cognitive function based on how fast they can search, scan, and process visual information. These scores are normalized to reflect a 1-100 percentile range. Higher scores indicate better performance.

CONTACTS AND LOCATIONS:
Overall Officials: Simon W Davis, PhD, Principal Investigator — Duke University; Andy Liu, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No